CLINICAL TRIAL: NCT04543539
Title: IN.PACT™ AV Access Post-Approval Study (PAS002)
Status: Active, not recruiting | Type: Observational
Sponsor: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: IN.PACT™ AV Access PAS002
Record Dates: First submitted 2020-09-02; First posted 2020-09-10 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-09

CONDITIONS: Arteriovenous Fistula; Arteriovenous Fistula Stenosis; Arteriovenous Fistula Occlusion; Fistula
MeSH Terms: conditions — Arteriovenous Fistula; Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- IN.PACT™ AV Access PAS Primary Cohort: The primary cohort consists of enrolled subjects treated with the IN.PACT™ AV DCB according to labeling requirements who meet the inclusion/exclusion criteria for the primary cohort.
  Interventions: Combination Product: IN.PACT™ AV Drug Coated Balloon (DCB) - Primary Cohort
- IN.PACT™ AV Access PAS Extended Cohort: The extended cohort consists of enrolled subjects who do not meet the eligibility criteria for the primary cohort and receive the IN.PACT™ AV DCB device for treatment of stenosis in the AV circuit.
  Interventions: Combination Product: IN.PACT™ AV Drug Coated Balloon (DCB) - Extended Cohort

INTERVENTIONS:
Combination Product: IN.PACT™ AV Drug Coated Balloon (DCB) - Primary Cohort — For the treatment of obstructive lesions up to 100 mm in length in the native arteriovenous dialysis fistulae with reference vessel diameters of 4 to 12 mm.
  Groups: IN.PACT™ AV Access PAS Primary Cohort
Combination Product: IN.PACT™ AV Drug Coated Balloon (DCB) - Extended Cohort — For treatment of stenosis in the AV circuit
  Groups: IN.PACT™ AV Access PAS Extended Cohort

SUMMARY:
Long-term safety will be summarized

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the long-term safety of the IN.PACT™ AV Access Drug Coated Balloon (DCB) for treatment of subjects presenting with de novo or non-stented restenotic obstructive lesion of native arteriovenous dialysis fistulae (AVF) in the upper extremity. Patients will be followed for five years. The IN.PACT™ AV Access PAS 002 is required by the Food and Drug Administration (FDA) as a condition of product approval. This study is conducted within Medtronic's post market surveillance platform.

ELIGIBILITY:
Primary Cohort Inclusion Criteria:

* Patient is ≥ 21 years of age
* Patient has a mature native AV fistula created ≥ 60 days prior to the index procedure
* Patient has a de novo and/or non-stented restenotic lesion located between the arteriovenous anastomosis and axillosubclavian junction
* Patient has a target lesion or a tandem lesion that is ≤ 100 mm in length (by visual estimate) Note: Tandem lesions may be included provided they meet all of the following criteria: a. Separated by a gap of ≤ 30 mm (3 cm), b. Total combined lesion length, including 30 mm gap, ≤ 100 mm, c. Able to be treated as a single lesion
* Patient has a target vessel diameter of 4.0 - 12.0 mm (by visual estimate)
* Patient underwent successful crossing of the target lesion with the guide wire and pre-dilatation with a PTA balloon defined as: Residual stenosis of ≤ 30% AND Absence of a flow limiting dissection or perforation AND No extravasation requiring treatment

Primary Cohort Exclusion Criteria:

* Women who are breastfeeding, pregnant, or are intending to become pregnant, or men intending to father children
* Patient is receiving immunosuppressive therapy
* Patient has an infected AV access or systemic infection
* Patient with hemodynamically significant central venous stenoses that cannot be successfully treated prior to treatment of the target lesion
* Patient with target lesion located central to the axillosubclavian junction
* Patient has significant arterial inflow lesion requiring treatment more than 2 cm upstream from the anastomosis in the AV access
* Patient has presence of pseudoaneurysm or aneurysm requiring treatment at the lesion site
* Target lesion is located within a bare metal or covered stent
* Patients with known allergies or sensitivities to paclitaxel
* Patient with known contraindication, including allergic reaction, or sensitivity to contrast material that cannot be adequately pre-treated
* Patient who cannot receive recommended antiplatelet and/or anticoagulant therapy
* Patient is enrolled in another investigational drug, device, or biologic study and has not completed the primary endpoint, or was previously enrolled in this study
* Patient has a co-morbid condition that, in the judgment of the Investigator, may cause him/her to be non-compliant with the protocol or confound the data interpretation
* Patient has an active COVID-19 infection with ongoing sequela at enrollment or hospitalization for treatment of COVID-19

Inclusion Criteria for Extended Cohort:

* Patient is ≥ 21 years of age

Exclusion Criteria for Extended Cohort:

* Patient has an active COVID-19 infection with ongoing sequela at enrollment or hospitalization for treatment of COVID-19

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes patients that will have an angioplasty with the IN.PACT™ AV Paclitaxel-Coated PTA Balloon Catheter (IN.PACT™ AV DCB).
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2025-06-03 (Actual); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Infection and Infestations Serious Adverse Events | Through 12 months post-index procedure
  Demonstrate Infection and Infestations Serious Adverse Events, including pneumonia, meets the performance goal of 30% in the primary cohort.

SECONDARY OUTCOMES:
Mortality Rate | Through 1, 2, 3, 4, and 5 years post-index procedure
  Determine mortality rate

OTHER OUTCOMES:
Extended Cohort - Characterize Infections and Infestations Serious Adverse Events | Through 1-year and all-cause mortality through 5-years post-index procedure
  Characterize infections and infestations Serious Adverse Events, including pneumonia.

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Cedars-Sinai Heart Institute, Los Angeles, California
  - Stanford University Medical Center, Stanford, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - Medstar Washington Hospital, Washington D.C., District of Columbia
  - NCH Healthcare System, Naples, Florida
  - Coastal Vascular and Interventional, Pensacola, Florida
  - University of Iowa, Iowa City, Iowa
  - University of Michigan Health System - University Hospital, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Holy Name Medical Center, Teaneck, New Jersey
  - Albany Medical College, Albany, New York
  - The Mount Sinai Hospital, New York, New York
  - Staten Island University Hospital, Staten Island, New York
  - FirstHealth of the Carolinas, Pinehurst, North Carolina
  - Oregon Health & Science University Hospital, Portland, Oregon
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - MUSC Health Dialysis Access Institute, Orangeburg, South Carolina
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - University of Virginia Medical Center, Charlottesville, Virginia
  - University of Wisconsin-Madison - Meriter Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No